CLINICAL TRIAL: NCT04647955
Title: Validation of a Questionnaire for Symptom Assessment in Postprandial Distress Syndrome (Functional Dyspepsia)
Brief Title: Functional Dyspepsia: Validation of a Questionnaire for Symptom Assessment in FD PDS Subgroup
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: LPDSItopride
Record Dates: First submitted 2020-11-16; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Functional Dyspepsia; Postprandial Fullness Syndrome
MeSH Terms: interventions — itopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itopride (Experimental): Oral dose of itopride 100 mg three times daily before the meal for 8 weeks
  Interventions: Drug: Itopride
- Placebo (Placebo Comparator): Oral dose of placebo three times daily before the meal for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itopride — Itopride is a D2 antagonist and cholinesterase inhibitor with prokinetic effects on gastric motility used to treat functional dyspepsia. Patients were treated for 8 weeks.
  Arms: Itopride
Drug: Placebo — Patients were treated for 8 weeks.
  Arms: Placebo

SUMMARY:
Fuctional dyspepsia is defined as the presence of symptoms thought to originate from the gastroduodenum, in the absence of any structural or metabolic disease that is likely to explain these symptoms. To facilitate its diagnostic and therapeutic approach, the Rome consensus proposed to distinguish 2 subgroups: postprandial distress syndrome (PDS), is characterized by meal-related symptoms such as early satiation and postprandial fullness. At present, no validated instrument is available for the assessment of the symptom responsiveness in patients suffering from PDS. To develop a new PRO questionnaire, we have previously conducted focus group sessions and cognitive interviews in PDS patients to identify all relevant symptom items that characterize PDS. In this study we aim to validate the provisional Leuven Postprandial Distress Scale (LPDS) through the assessment of its consistency, reliability and ability to detect change in the framework of a controlled treatment trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PDS diagnosis as per Rome III by Rome III questionnaire (see appendix 1B)
* Patients must provide witnessed written informed consent prior to any study procedures being performed
* Patients aged between 18 and 70 years inclusive
* Male or female patients
* Patients who are capable to understand the study and the questionnaires, and to comply with the study requirements

Exclusion Criteria:

* Patients with any condition which, in the opinion of the investigator, makes the patient unsuitable for entry into the study
* Patients with an active major psychiatric condition (depression, anxiety disorder, alcohol or substance abuse). Patients who are taking a stable dose of a single antidepressant (with the exception of amitryptiline) during the last 3 months are eligible.
* Females who are pregnant or lactating.
* Patients who are H. Pylori positive or patients who received treatment for HP eradication during the last 3 months.
* Patients suffering from diabetes type 1 or type 2.
* Patients taking medication for functional dyspepsia will need a wash-out period of 2 weeks before they can be screened
* Patients with known hypersensitivity to gastroprokinetic drugs.
* Patients with confirmed gastro-intestinal disease.
* Patients with former digestive surgery affecting upper gut motility.
* Patients affected by concomitant disease responsible for digestive symptoms
* Patients presenting with predominant symptoms of irritable bowel syndrome (IBS)
* Patients presenting symptoms of EPS several times a week according to Rome III questionnaire
* Patients presenting daily symptoms of CIN on Rome III questionnaire
* Patients presenting vomiting more than one day a month.
* Patients presenting daily symptoms of Excessive belching according to Rome III questionnaire
* Patients presenting predominant GERD according to GERD questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Validation of LPDS questionnaire | 8 weeks
  Responsiveness of LPDS

SECONDARY OUTCOMES:
Percentage of subject that improved after treatment with itopride based on the LPDS validated questionnaire | 8 weeks
  Percentage of subjects that show a decrease of at least 0.5 in the LPDS score at the end of the treatment. We calculated the number of patients that reached the LPDS MCID (≥0.5) and at a higher response threshold (≥0.7) and differences between proportions were analysed with the Chi-squared test.
Efficacy of itopride compared to baseline based on the LPDS validated questionnaire | 8 weeks
  Improvement of dyspepsia symptoms at the end of the treatment compared to baseline. Within each treatment arm, the change from baseline to week 8 of treatment in quantitative measures was evaluated by mixed models.
Efficacy of itopride compared to baseline in the dyspepsia subgroups on based on the LPDS validated questionnaire | 8 weeks
  Improvement of dyspepsia symptoms at the end of the treatment compared to baseline. Within each treatment arm, the change from baseline to week 8 of treatment in quantitative measures was evaluated by mixed models.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carbone F, Vandenberghe A, Holvoet L, Piessevaux H, Arts J, Caenepeel P, Staessen D, Vergauwe P, Maldague P, De Ronde T, Wuestenberghs F, Lamy V, Lefebvre V, Latour P, Vanuytsel T, Jones M, Tack J. A double-blind randomized, multicenter, placebo-controlled study of itopride in functional dyspepsia postprandial distress syndrome. Neurogastroenterol Motil. 2022 Aug;34(8):e14337. doi: 10.1111/nmo.14337. Epub 2022 Mar 31. PMID 35357058